CLINICAL TRIAL: NCT04374695
Title: Association Between Hypertension, Renin-Angiotensin-Aldosterone System Inhibitors and COVID-19
Brief Title: Renin-Angiotensin-Aldosterone System Inhibitors, Hypertension, and COVID-19
Acronym: COVHYP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Versailles Hospital (Other)
Collaborators: Bernard LIVAREK, MD, Cardiology department, Versailles Hospital (Unknown); Jean-Paul BERESSI, MD, Department of diabetology, Versailles Hospital (Unknown); Mehrsa KOUKABI FRADELIZZI, MD, Emergency department, Versailles Hospital (Unknown); Floriane GILLES, MD, Cardiology department, Versailles Hospital (Unknown); Alisson BERTRAND, Cardiology department, Versailles Hospital (Unknown); Marie DE TOURNEMIRE, Cardiology department, Versailles Hospital (Unknown); Victorien MONGUILLON, Cardiology department, Versailles Hospital (Unknown); Maeva PASQUALINI, Cardiology department, Versailles Hospital (Unknown); Alix PREVOT, Cardiology department, Versailles Hospital (Unknown); Guillaume ROGER, Cardiology department, Versailles Hospital (Unknown); Joseph SABA, Cardiology department, Versailles Hospital (Unknown); Joséphine SOLTANI, Cardiology department, Versailles Hospital (Unknown); Jean-François PROST, Cardiology department, Versailles Hospital (Unknown); Cécile LAUREANA, Department of medical information, Versailles Hospital (Unknown)
Responsible Party: Principal Investigator, Jean-Louis GEORGES, MD, MPH, FESC, Versailles Hospital
Other Study IDs: P20/11_COVHYP
Record Dates: First submitted 2020-05-03; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: COVID-19; Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Blockers; Renin-Angiotensin System; Hypertension; Observational Study
MeSH Terms: conditions — COVID-19; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with COVID-19: Patients with positive RT-PCR for SARS-CoV-2, and patients with négative RT-PCR for SARS-CoV-2 but clinical presentation highly suggestive of COVID-19, and typical COVID-19 abnormalities on chest CT-Scan.
- patients without COVID-19: Patients with négative RT-PCR for SARS-CoV-2 and chest CT-Scan or chest X-ray not suggestive of COVID-19

SUMMARY:
Background. Angiotensing converting enzyme type 2 (ACE2), a key enzyme of the renin-angiotensin-aldosterone system (RAAS), is the receptor of SARS-CoV-2 for cell entry into lungs. Because ACE2 may be modulated by RAAS inhibitors, such as angiotensin converting enzyme inhibitors (ACEi) and angiotensin II receptor blockers (ARBs), there is concern that patients treated with ACEi and ARBs may be at higher risk for COVID-19 infection and severity.

Aim. To analyze the associations between COVID-19 and hypertension, and treatments with ACEi and ARBs.

Methods. In this retrospective observational study, consecutive patients hospitalized for suspected COVID-19 pneumonia will be divided into 2 groups, whether or not COVID-19 is confirmed. The two groups will be compared for baseline characteristics, mainly prior treatment with ACEi and ARBs, and clinical outcome at 1-month follow-up.

The main hypothesis is that ACEi and ARBs, which interact differently with ACE2, may have different relationships with COVID-19 infection or severity.

DETAILED DESCRIPTION:
The coronavirus disease 2019 (Covid-19) pandemic is currently the main challenge facing healthcare providers. Data are lacking to guide clinical decision.

The renin-angiotensin-aldosterone system (RAAS) is a key process in cardiology. Its inhibition using angiotensin-converting enzyme inhibitors (ACEi) and angiotensin II type 1-receptor blockers (ARBs) is a cornerstone of the long-term management of arterial hypertension, heart failure and acute coronary syndrome. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) uses the angiotensin-converting enzyme 2 (ACE2) as a cellular entry receptor. ACE2 is part of the RAAS and is likely to be modulated by the use of ACEi and ARBs. Therefore, there is concern that patients who are treated with ACEi and ARBs may be at higher risk for Covid-19 infection.

However, little is known regarding how ACEi and ARBs could affect Covid-19 infection and severity. First, ACE2 may have a protective effect against lung injury because it degrades angiotensin II to angiotensin-(1-7). Second, the effect of RAAS inhibition on ACE2 expression has been poorly studied in humans. Third, ACE inhibitors and ARB have different effect on the RAAS and therefore their interaction with Covid-19 may differ.

The COVHYP study is designed to address part of these issues. This is an analytical retrospective observational study that will collect and analyze data regarding patients hospitalized with suspected Covid-19. We planned to screen for inclusion all consecutive patients referred form 10/03/2020 to 15/04/2020 to the emergency department of the Versailles Hospital, a tertiary center located in greater Paris area - one of the region most affected by Covid-19 in France through this period. The inclusion criteria are as follows: 1) Clinical presentation suggestive of COVID-19 pneumonia, at least fever or influenza-like syndrome AND cough or dyspnea; and 2) Test of the presence of SARS-CoV-2 RNA by RT-PCR in nasopharyngeal or sputum samples. Two groups of patients will be defined, those with confirmed Covid-19 pneumonia, and those without Covid-19. Hospital data will gathered, and patients or relatives will be contacted by phone for a one-month follow-up. We will compare baseline characteristics of patients, especially the previous treatment by ACEi or ARBs, in the two groups of patients, and evaluate whether these characteristics can be associated with diagnosis of SARS-CoV-2 infection and severity.

We hope that this study will provide a better understanding of the effect of RAAS inhibitors on Covid-19 pneumonia and its severity.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or more than 18;
* Symptoms suggestive of Covid-19 pneumonia. At least : fever > 38°C or influenza-like illness (asthenia, myalgia, chills, muscular aches, …) AND cough or dyspnea;
* Hospitalization required on clinical criteria including: oxygen saturation <96% without oxygen support, respiratory frequency > 25 per minute, hemodynamic instability, medical history or comorbidities known at high risk for Covid-19 (chronic heart disease, congestive heart failure, chronic bronchopulmonary disease, diabetes mellitus, age>70, history of cancer, immunosuppression, …);
* Covid-19 confirmation test performed (RT-PCR).

Exclusion Criteria:

* Age < 18
* Refusal to participate in the study
* detainee or prisoner
* Protected adult uncapable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients presenting to the Centre hospitalier de Versailles emergency department from 2020 March 10th to April, 15th with clinical symptoms suggestive of COVID-19, who fulfilled the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Prior treatment by ACEi | at admission to hospital
  Prevalence of a previous treatment by angiotensin converting enzyme inhibitors in patients with and without confirmed Covid-19 pneumonia.
Prior treatment by ARB | at admission to hospital
  Prevalence of a previous treatment by angiotensin II type 1-receptor blockers in patients with and without confirmed Covid-19 pneumonia.

SECONDARY OUTCOMES:
Baseline characteristics and comorbidities | at admission to hospital
  Association between COVID-19 infection status and other baseline characteristics and comorbidities (age, sex, history of hypertension, chronic heart disease, diabetes mellitus, COPD, asthma, obesity, allergies)
Major Clinical Adverse Events | One month follow-up
  Association between previous treatment by ACEi and ARBs and clinical course of COVID-19 (one-month mortality, hospitalization in intensive care unit, duration of hospital stay, early discharge to home)

IPD SHARING:
Plan to Share IPD: Undecided